CLINICAL TRIAL: NCT04011995
Title: Effects of Intermittent Caloric Restriction in Youth With Cardiometabolic Risk: a Randomized Controlled Pilot Study
Brief Title: Effects of Intermittent Caloric Restriction in Youth With Cardiometabolic Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Weili Yan, Professor, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICR_2019_2.0
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Overweight; Obesity; Cardiometabolic Risk
Keywords: Intermittent caloric restriction; Children; Youth
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent caloric restriction (Experimental)
  Interventions: Behavioral: Intermittent caloric restriction; Behavioral: Health education on reducing the cardiometabolic risk
- Low carbohydrate diet (Active Comparator)
  Interventions: Behavioral: Low carbohydrate diet; Behavioral: Health education on reducing the cardiometabolic risk

INTERVENTIONS:
Behavioral: Intermittent caloric restriction — The intervention is based on the 5:2 diet, which involves caloric restriction for 2 days (consecutive or nonconsecutive, 600kcal/d for male and 500kcal/d for female) per week and unrestricted eating during the other 5 days of the week.
  Total trial duration is one month consisting of a 14-day intervention phase and a 14-day self-maintenance phase. During the maintenance phase, two follow-up electronic questionnaires were conducted.
  Other Names: Intermittent fasting
  Arms: Intermittent caloric restriction
Behavioral: Low carbohydrate diet — During the 14-day intervention period, the subjects receive 7 days (consecutive or nonconsecutive) of low carbohydrate diet intervention. Carbohydrate intake of low-carbohydrate diet should be controlled as ≤ 50g per day.
  Total trial duration is one month consisting of a 14-day intervention phase and a 14-day self-maintenance phase. During the maintenance phase, two follow-up electronic questionnaires were conducted.
  Arms: Low carbohydrate diet
Behavioral: Health education on reducing the cardiometabolic risk — Health education is conducted once a week during 14-day dietary intervention for all subjects. Health education including the understanding of cardiovascular disease, how to determine the cardiometabolic risk level, and the lifestyle intervention as caloric restriction and increased physical activity to promote health.

SUMMARY:
This is a randomized controlled pilot study to evaluate the effects of intermittent caloric restriction compared with low carbohydrate diet in youth with cardiometabolic risk.

DETAILED DESCRIPTION:
The National China Health and Nutrition Survey revealed that 42% of overweight children had at least one cardiovascular metabolic risk, such as hyperglycaemia, dyslipidemia or hypertension. Non-pharmaceutical life style modifications are the recommended intervention to these subjects, including caloric restriction and increased physical activity. However, the problems of poor compliance and metabolic adaptation are well known. Evidences from a number studies in rodent models and human indicated that intermittent caloric restriction (ICR) may stimulate series reactions in human body, including improvement of insulin sensitivity, blood pressure, oxidative stress and inflammation, and may be easier to follow. Evidence from larger human studies is strongly encouraged, while the effects, safety and adherence in chidren and youth need to be studied.

This study is a randomized controlled trial of intermittent caloric restriction versus low carbohydrate diet in youth with cardiometabolic risk over one month period. The intervention is based on the 5:2 diet, which involves caloric restriction for 2 days (consecutive or nonconsecutive, 600kcal/d for male and 500kcal/d for female) per week and unrestricted eating during the other 5 days of the week. For control group, the subjects receive 7 days (consecutive or nonconsecutive) of low carbohydrate diet intervention during the 14-day intervention period,. Carbohydrate intake of low-carbohydrate diet should be controlled as ≤ 50g per day. Total trial duration is one month consisting of a 14-day intervention phase and a 14-day self-maintenance phase. During the maintenance phase, two follow-up electronic questionnaires were conducted.

The study aim to explore effects of the dietary interventions on cardiometabolic markers, inflammatory reaction, oxidative stress and gut microbiome in youth with cardiometabolic risk.

ELIGIBILITY:
Inclusion Criteria:

Have at least one of the following cardiometabolic abnormalities:

1. Overweight or obesity (central obesity or general obesity)
2. Prediabetes: impaired fasting glucose (IFG) and/or impaired glucose tolerance (IGT)
3. Dyslipidemia
4. Elevated blood pressure

Criteria for cardiometabolic abnormalities:

1. Overweight or obesity

   For subjects (9 ≤ age ≤ 18 years) :

   • General obesity: Body mass index higher than the 85th percentile for overweight and the 90th percentile for obesity, based on the references for screening overweight and obesity in Chinese children and adolescents.

   • Central obesity: Waist circumference higher than the 90th percentile of the age and gender-specific reference for screening cardiovascular risk factors in Chinese children and adolescents.

   For subjects ( 19 ≤ age ≤ 30 years) :

   • General obesity: Body mass index between 24.0 and 27.9 kg/m2 for overweight and ≥28 kg/m2 for obesity.

   • Central obesity: Waist circumference ≥85cm for men and ≥80cm for female. Based on recommendation of overweight and obesity in Chinese adults.
2. Prediabetes:

   With IFG and/or IGT. IFG: fasting glucose from 5.6 to 6.9 mmol/L; IGT: 2-h glucose in the 75g oral glucose tolerance test from 7.8 to 11.0 mmol/L.

   Based on recommendation of American Diabetes Association.
3. Dyslipidemia:

   For subjects (9 ≤ age ≤ 18 years) :

   Triglycerides of ≥1.70 mmol/L or total cholesterol of ≥5.18 mmol/L or lowdensity lipoprotein cholesterol ≥3.37 mmol/L or highdensity lipoprotein cholesterol of ≤1.04 mmol/L. Based on recommendation in Chinese children and adolescents.

   For subjects ( 19 ≤ age ≤ 30 years) :

   Triglycerides of ≥1.7 mmol/L or total cholesterol of ≥5.2 mmol/L or lowdensity lipoprotein cholesterol ≥3.4 mmol/L or highdensity lipoprotein cholesterol of ≤1.0 mmol/L. Based on guideline for the management of dyslipidemia in Chinese adults.
4. Elevated blood pressure:

For subjects (9 ≤ age ≤ 18 years) :

Blood pressure higher than the 90th percentile of blood pressure age and gender-specific reference standards for Chinese children and adolescents, or blood pressure >120/80 mmHg.

For subjects ( 19 ≤ age ≤ 30 years) :

Systolic blood pressure≥120 mmHg and/or diastolic blood pressure ≥80 mmHg. Based on Chinese guidelines for the management of hypertension.

Exclusion Criteria:

1. Diagnosis of severe diseases such as cardiac insufficiency, severe malnutrition or immunodeficiency.
2. History of bariatric surgery.
3. Use of antiobesity drugs or supplements.

Ages: 9 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Reversal of cardiometabolic abnormalities | From the baseline (the first day of the intervention phase) to the 14th day of the intervention phase.
  The primary outcome is a composite outcome that will be measured by combining multiple reverse outcomes of the following cardiometabolic abnormalities: (1) overweight or obesity, (2) prediabetes, (3) hyperlipidemia and (4) elevated blood pressure. It is defined as occurring if any cardiometabolic abnormality has a reversal outcome at the 14th day of dietary intervention phase.
  Reversal of cardiometabolic abnormalities is defined as:
  At the 14th day of dietary intervention phase, at least one of the following indicators changed from abnormal at baseline to normal: overweight, obesity, prediabetes, hyperlipidemia and elevated blood pressure.
  (The reversal of overweight or obesity is defined according to reference[1, 2]: For subject with general obesity at baseline: weight loss of 1.5 kg after intervention; For subject with central obesity at baseline: waist circumference reduction of 1.5 cm after intervention.)

SECONDARY OUTCOMES:
Change in insulin | From the baseline (the first day of the intervention phase) to the 14th day of the intervention phase.
  Serum from fasting blood sample is used for measurement of insulin.
Change in insulin-like growth factor-1 | From the baseline (the first day of the intervention phase) to the 14th day of the intervention phase.
  Fasting blood sample for measurement of insulin-like growth factor-1.
Change in mean blood glucose | From the baseline (the first day of the intervention phase) to the 14th day of the intervention phase.
  Measured by a blood glucose monitor for 24-hour glucose monitoring during the 14-day intervention phase.
Change in gut microbial compositions | From the baseline (the first day of the intervention phase) to the 14th day of the intervention phase.
  Stool sample of subject is used for measurement of gut microbial compositions.
Change in body weight | From the baseline (the first day of the intervention phase) to the 14th day of the intervention phase.
  Body weight is measured according to the Physical Fitness and Health Surveillance of Chinese School Students by trained, certified study staff. It is measured to the nearest 0.1 kg.
Change in body weight | From the baseline (the first day of the intervention phase) to the 14th day of the self-maintenance phase.
  Body weight is measured by subject and reported by electronic questionnaire. It is measured to the nearest 0.1 kg.
Change in waist circumference | From the baseline (the first day of the intervention phase) to the 14th day of the intervention phase.
  Waist circumference is measured to the nearest 0.1 cm using a constant tension tape around the waist at 1 cm below the navel as the subject exhaled. It is calculated as the average value of two measurements.
Change in waist circumference | From the baseline (the first day of the intervention phase) to the 14th day of the self-maintenance phase.
  Waist circumference is measured by subject and reported by electronic questionnaire. It is measured to the nearest 0.1 cm using a constant tension tape around the waist at 1 cm below the navel as the subject exhaled. It is calculated as the average value of two measurements.
Dietary energy intake | From the baseline (the first day of the intervention phase) to the 14th day of the intervention phase.
  Daily dietary energy intake (kcals/day) is calculated by researchers using food weighing photos of the subject.
Self-reported dietary adherence | At the 14th day of the self-maintenance phase.
  Adherence to diet will be assessed with a electronic questionnaire in the self-maintenance phase.
Change in monocyte chemoattractant protein-1 (MCP-1) | From the baseline (the first day of the intervention phase) to the 14th day of the intervention phase.
  MCP-1 will be measured by enzyme-linked immunosorbent assays (R&D Systems, Inc. USA), using fasting serum samples at baseline and 14 days after intervention.
Change in free fatty acid (FFA) | From the baseline (the first day of the intervention phase) to the 14th day of the intervention phase.
  FFA will be measured by enzyme-linked immunosorbent assays (R&D Systems, Inc. USA), using fasting serum samples at baseline and 14 days after intervention.
Change in fibroblast growth factor 21 (FGF-21) | From the baseline (the first day of the intervention phase) to the 14th day of the intervention phase.
  FGF-21 will be measured by enzyme-linked immunosorbent assays (R&D Systems, Inc. USA), using fasting serum samples at baseline and 14 days after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

REFERENCES:
- [Background] Harvie MN, Pegington M, Mattson MP, Frystyk J, Dillon B, Evans G, Cuzick J, Jebb SA, Martin B, Cutler RG, Son TG, Maudsley S, Carlson OD, Egan JM, Flyvbjerg A, Howell A. The effects of intermittent or continuous energy restriction on weight loss and metabolic disease risk markers: a randomized trial in young overweight women. Int J Obes (Lond). 2011 May;35(5):714-27. doi: 10.1038/ijo.2010.171. Epub 2010 Oct 5. PMID 20921964
- [Background] Arnason TG, Bowen MW, Mansell KD. Effects of intermittent fasting on health markers in those with type 2 diabetes: A pilot study. World J Diabetes. 2017 Apr 15;8(4):154-164. doi: 10.4239/wjd.v8.i4.154. PMID 28465792
- [Derived] Dou Y, Jiang Y, Chen X, Zhang Y, Wang Y, Chen H, He W, Yan W. Intermittent dietary carbohydrate restriction versus calorie restriction and cardiometabolic profiles: A randomized trial. Obesity (Silver Spring). 2023 Sep;31(9):2260-2271. doi: 10.1002/oby.23855. Epub 2023 Aug 7. PMID 37545298

DOCUMENTS (2):
  • Study Protocol (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT04011995/Prot_001.pdf
  • Statistical Analysis Plan (2019-09-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT04011995/SAP_000.pdf